CLINICAL TRIAL: NCT06848504
Title: Implementing MedSMA℞T Families in the Emergency Department Setting: A Game-based Approach for Improving Opioid Safety Among Adolescents and Parents
Brief Title: MedSMA℞T Mobile ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olufunmilola Abraham (Other)
Responsible Party: Sponsor-Investigator, Olufunmilola Abraham, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 98853; R18HS030202 (AHRQ)
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Opiate-Related Disorders; Opiate Use Disorder; Opioid
Keywords: Opioid Education; Opioid Use Disorder; Opiate-Related Disorders; Opiate; Opioid; Serious Game; Smartphone; Smartphone Game; Medication safety; Adolescent Health
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This group will receive the intervention of interest, MedSMA℞T Mobile, in addition to standard opioid-related counseling. MedSMA℞T Mobile is a serious game (intended to educate while entertaining) focused on opioid safety.
  Interventions: Behavioral: MedSMA℞T Mobile
- Control (No Intervention): This group will receive the standard opioid-related counseling that all patients receive when newly prescribed opioids in the emergency department.

INTERVENTIONS:
Behavioral: MedSMA℞T Mobile — MedSMA℞T Mobile is an innovative mobile digital health intervention that integrates technology-based learning to facilitate family communication and creation of a personalized Family Medication Safety Plan. The Family Medication Safety Plan (FMSP) is a tool for families to record important information about their medications and create a plan for safe use, storage, and disposal. Participants will play MedSMA℞T Mobile for up to 30 minutes at the first study visit.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if a new smartphone-based intervention can help with factors related to opioid misuse in parents and adolescent/early adult children. The main question it aims to answer is:

• Can this intervention improve knowledge of, and attitudes towards, opioid misuse over traditional opioid-related counseling alone?

Participants will, in addition to receiving opioid counseling:

* Join an online meeting with research staff to test the smartphone-based intervention
* Report demographic information
* Complete surveys about opioids
* Complete a family medication safety plan
* Complete surveys after 3, 6, and 9 months

ELIGIBILITY:
Inclusion Criteria:

* Adults who receive an opioid prescription from a study Emergency Department, AND
* who report having an adolescent, aged 12-18, living at home, AND
* who speak and understand English
* Each participant must have the ability to provide informed consent

Exclusion Criteria:

* Adults who do not receive an opioid prescription from a study Emergency Department AND/OR
* who do not have an adolescent, aged 12-18, living at home, AND/OR
* who do not speak or understand English
* Adults and/or adolescents who do not have the ability to provide informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Adolescent Opioid Safety and Learning (AOSL) scale score over 9 month study | Baseline, 3, 6, and 9 months.
  The fourth factor of the Adolescent Opioid Safety and Learning (AOSL) scale, Opioid Harm, measures understanding of negative social and professional effects of opioid misuse. Scores range from 3-15, where 3 indicates the lowest level of overall opioid harm awareness and 15 is the highest level.

SECONDARY OUTCOMES:
Change in Safe Opioid Storage Behaviour over 9 months | Baseline, 3, 6, and 9 months.
  This outcome contains 4 items from the Wisconsin Strategic Prevention Framework Partnerships for Success Community Survey - V02, comprised of yes/no questions. The minimum score for this scale is 0 (indicating least safe opioid storage behaviour) and the maximum is 4 (indicating most safe opioid storage behaviour).
Change in Opioid Disposal Behaviour over 9 months | Baseline, 3, 6, and 9 months.
  This outcome contains 6 items from the Wisconsin Strategic Prevention Framework Partnerships for Success Community Survey - V02, and includes yes/no questions. The minimum score for this scale is 0 (indicating least safe opioid disposal behaviour) and the maximum is 6 (indicating most safe opioid disposal behaviour).
Change in Medication Understanding and Use Self-Efficacy (MUSE) scale scores over 9 months | Baseline, 3, 6, and 9 months.
  This section covers the second factor, Learning About Medication, of the Medication Understanding and Use Self-Efficacy (MUSE) scale. This factor is comprised of 4 items, each scored 1-4. The minimum score is 4, and the maximum is 16. A score of 4 indicates lower understanding and self-efficacy in opioid use, whereas a score of 16 indicates highest level of understanding and self-efficacy in opioid use.
Change in Family Communication Behaviour Patterns over 9 months | Baseline, 3, 6, and 9 months.
  This includes both the parent and child versions of the 26-item, 2-factor scales. The first factor, Conversation orientation, contains 15 items. The second factor, Conformity orientation, contains 11 items. Items are scored from 1-5, where 1 is "Disagree Strongly" and 5 is "Agree Strongly". Scale scores are averages for the two scales, with each item contributing equally. The minimum and maximum average scores, therefore, cannot exceed 1 and 5, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilola Abraham, PhD, Principal Investigator — University of Kentucky College of Pharmacy
Locations (3):
- United States (3):
  - Swedish American Hospital, Rockford, Illinois
  - East Madison Hospital, Madison, Wisconsin
  - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No